CLINICAL TRIAL: NCT05238883
Title: A Phase 1a/1b, Open-Label, Multi-Center, Dose Escalation and Expansion Study of HFB200301 (TNFR2 Agonist Antibody) as a Single Agent and in Combination With Tislelizumab (Anti-PD-1 Antibody) in Adult Patients With Advanced Solid Tumors
Brief Title: A Study of HFB200301 as a Single Agent and in Combination With Tislelizumab in Adult Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HiFiBiO Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HFB-200301-01; 2021-006231-25 (EudraCT Number); 2024-511286-11-00 (EU CTIS Number)
Record Dates: First submitted 2021-12-16; First posted 2022-02-14 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Gastric Cancer; Renal Cell Carcinoma; Melanoma; Sarcoma; Testicular Germ Cell Tumor; Cervical Cancer; Mesothelioma; Non Small Cell Lung Cancer; Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Stomach Neoplasms; Carcinoma, Renal Cell; Melanoma; Sarcoma; Testicular Germ Cell Tumor; Uterine Cervical Neoplasms; Mesothelioma; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck | interventions — tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation - HFB200301 monotherapy (Experimental): Participants will be administered HFB200301 at dose levels 1-5 as an intravenous infusion to determine the Recommended Dose for Expansion (RDE).
  Interventions: Drug: HFB200301
- Dose Escalation - HFB200301 in combination with tislelizumab (Experimental): Participants will be administered HFB200301 at dose levels 1-4 in combination with one dose level of tislelizumab as an intravenous infusion to determine the combination Recommended Dose for Expansion (RDE).
  Interventions: Drug: HFB200301; Drug: Tislelizumab
- Dose Expansion - HFB200301 monotherapy (Experimental): Participants will be administered HFB200301 at monotherapy RDE as an intravenous infusion.
  Interventions: Drug: HFB200301
- Dose Expansion - HFB200301 in combination with tislelizumab (Experimental): Participations will be administered HFB200301 in combination with tislelizumab at combination RDE as an intravenous infusion.
  Interventions: Drug: HFB200301; Drug: Tislelizumab

INTERVENTIONS:
Drug: HFB200301 — Participants will be administered HFB200301 as described in the experimental arm.
Drug: Tislelizumab — Participants will be administered tislelizumab as described in the experimental arm.
  Other Names: BGB-A317
  Arms: Dose Escalation - HFB200301 in combination with tislelizumab; Dose Expansion - HFB200301 in combination with tislelizumab

SUMMARY:
The purpose of this study is to test the safety and tolerability of HFB200301 as a single agent and in combination with tislelizumab in patients with advanced cancers. There are two parts in this study. During the escalation part, groups of participants will receive increasing doses of HFB200301 as a monotherapy or in combination with tislelizumab until a safe and tolerable dose of HFB200301 as a single agent or combination therapy is determined. During the expansion part, participants will take the dose of HFB200301 as a monotherapy or in combination with tislelizumab that was determined from the escalation part of the study and will be assigned to a group based on the type of cancer the participants have.

DETAILED DESCRIPTION:
This is a Phase 1a/1b, first in human, open-label, dose escalation and expansion study in adults with advanced cancers. The study will comprise of

1. A Screening Period
2. A Treatment Period during which participants will receive the study drug on the first day of each cycle
3. A Follow-up Period

ELIGIBILITY:
Inclusion Criteria:

* Previously received the following lines of systemic therapy for the advanced/metastatic disease:

  * Gastric cancer: at least 2 lines of therapy
  * Renal cell carcinoma: at least 2 lines of therapy
  * Melanoma:

    * BRAF V600E mutant: must have received at least 2 lines of therapy
    * BRAF V600E wild type: must have received at least 1 line of therapy
  * Sarcoma: at least 1 line of therapy
  * Testicular germ cell tumor: at least 2 lines of therapy
  * Cervical cancer: at least 2 lines of therapy
  * Mesothelioma: at least 2 lines of therapy
  * Non-small cell lung cancer: at least 2 lines of therapy
  * Head and neck squamous cell carcinoma: at least 2 lines of therapy
* Suitable site to biopsy at pre-treatment and on-treatment
* Measurable disease as determined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or modified RECIST (mRECIST) for mesothelioma
* Eastern Cooperative Oncology Group performance status of 0 or 1

Exclusion Criteria:

* Systemic anti-cancer therapy within 2 weeks prior to start of study drug or within 4 weeks for immune-oncologic therapy
* For soft tissue sarcoma and testicular germ cell tumor patients only: prior immune therapy
* Therapeutic radiation therapy within the past 2 weeks
* Prior exposure to agents targeting the Tumor Necrosis Factor Receptor type 2 (TNFR2) receptor
* Active autoimmune disease requiring systemic treatment in the previous 2 years
* Systemic steroid therapy (>10 mg/day of prednisone or equivalent) or any immune suppressive therapy ≤ 14 days before first dose
* Persisting toxicity of ≥Grade 2 (≥Grade 1 for diarrhea) relating to prior anti cancer therapy with the following exceptions:

  * All grades of alopecia are acceptable
  * Endocrine dysfunction on replacement therapy is acceptable
* Severe or unstable medical condition, including uncontrolled diabetes, coagulopathy, or unstable psychiatric condition
* Major surgery within 4 weeks of the first dose of study drug
* History or presence of drug or non-drug induced interstitial lung disease or pneumonitis ≥Grade 2. For combination only: non-small cell lung cancer patients, mesothelioma or patients with significantly impaired pulmonary function or who require supplemental oxygen at baseline must undergo an assessment of pulmonary function at screening
* History of allergic reactions, immune related reactions, or cytokine release syndrome (CRS) attributed to compounds of similar chemical or biologic composition to monoclonal antibodies or any excipient of HFB200301
* Using sensitive substrates of major cytochrome P450 (CYP450) enzymes
* Known active malignancy, with the exception of the specific cancer under investigation in this trial, that required treatment within the previous 2 years
* For combination only:

  * Prior randomization in a tislelizumab study regardless of the treatment arm, until the primary and key secondary endpoints of the study have read out
  * Hypersensitivity to tislelizumab or any of its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs), serious AEs (SAEs), dose-limiting toxicities (DLTs), and tolerability (dose interruptions, reductions, and dose intensity) | assessed up to 3 years
To determine a Recommended Phase 2 Dose (RP2D) during Dose Expansion | assessed up to 3 years

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | assessed up to 3 years
Disease Control Rate (DCR) | assessed up to 3 years
Duration of Response (DOR) | assessed up to 3 years
Progression Free Survival (PFS) | assessed up to 3 years
Maximum serum concentration (Cmax) | average of 3 years
Terminal half-life (T1/2) | average of 3 years
Area under the concentration versus time curve (AUC) | average of 3 years
Serum concentration for measurement of anti-HFB200301 antibodies | average of 3 years
To assess the pharmacodynamic (PD) effects of HFB200301 as a single agent and in combination | average of 3 years
  Percent change in immunologic changes to immune cells

CONTACTS AND LOCATIONS:
Locations (10):
- United States (7):
  - Mayo Clinic, Scottsdale, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas
  - NEXT Virginia Cancer Specialists, Fairfax, Virginia
- Spain (3):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia

REFERENCES:
- [Derived] Gao Z, Zhang Q, Chen H, Chen J, Kang J, Yu H, Song Y, Zhang X. TNFR2 promotes pancreatic cancer proliferation, migration, and invasion via the NF-kappaB signaling pathway. Aging (Albany NY). 2023 Aug 16;15(16):8013-8025. doi: 10.18632/aging.204941. Epub 2023 Aug 16. PMID 37589506